CLINICAL TRIAL: NCT02558192
Title: Administration of a Lactobacillus GG and Vitamins Containing Mixture is Effective in Preventing Nosocomial Infection in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alfredo Guarino, Full Professor of Pediatrics, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IN001
Record Dates: First submitted 2015-04-13; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Nosocomial Infection
Keywords: LGG; Probiotics; nosocomial infection prevention; pediatrics
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Vials containing 3 x 10^9 Colony Forming Units of LGG, vitamins ( B and C) and zinc
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus GG
- Placebo (Placebo Comparator): Vials containing water, maltodextrin, magnesium stearate, potassium sorbate, sodium benzoate, citric acid, fructose, flavor.
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: Lactobacillus Rhamnosus GG — 1 vials q12 for 15 days
  Other Names: LGG
  Arms: Probiotics
Dietary Supplement: PLACEBO — 1 vials q12 for 15 days
  Arms: Placebo

SUMMARY:
Nosocomial infections are infections that occur from the time of 'entry in the hospital up to 48h after discharge. In most developed countries, the incidence of nosocomial infections in children is between 5% and 44% with the predominance of respiratory infections and gastrointestinal infections. Nosocomial infections prolong the time of hospital stay, reduce the effectiveness of treatment, significantly increasing hospital costs. Current measures for prevention of nosocomial infections in pediatrics, such as vaccinations and compliance with sanitary regulations, are not fully effective. Therefore it is necessary a deepening of the possible methods of prevention, between which has been already tested the use of probiotics such as Lactobacillus GG. A recent RCCT, which provided for the administration of LGG against placebo, noted a significant reduction in the risk of gastrointestinal infections and respiratory infections in hospitalized children treated with LGG, compared with patients who received placebo. There are also evidence which demonstrate a potential role zinc in reducing the incidence of respiratory infections is that bowel. We thought, therefore, to perform a multicenter randomized controlled trial with the aim to evaluate the role of a complex containing LGG, vitamins and zinc in the prevention of nosocomial gastrointestinal and respiratory tract infections in pediatric wards.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 3 months and 5 years
* Children admitted to a pediatric ward

Exclusion Criteria:

* Children with chronic diseases of the respiratory , gastrointestinal , renal system;
* Children with malformations of the cardiovascular system ;
* Children with immune deficiencies ;
* Infants born preterm ( gestational age < 37 weeks ) ;
* Children with congenital metabolic diseases ;
* Children Who received probiotics before enrollment ( up to 7 days before hospitalization)

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Study the incidence of nosocomial gastrointestinal infection | After 15 days of treatment
Study the incidence of nosocomial URTI | After 15 days of treatment

SECONDARY OUTCOMES:
Days of hospitalization | After 3 months from the enrollment
The incidence of gastrointestinal and respiratory infection during the 3 month follow-up period | After 3 months from the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Guarino, MD, Principal Investigator — Univesità degli Studi di Napoli "Federico II"
Locations (1):
- University of Naples "Federico II", Naples, Naples, Italy

REFERENCES:
- [Background] Hojsak I, Abdovic S, Szajewska H, Milosevic M, Krznaric Z, Kolacek S. Lactobacillus GG in the prevention of nosocomial gastrointestinal and respiratory tract infections. Pediatrics. 2010 May;125(5):e1171-7. doi: 10.1542/peds.2009-2568. Epub 2010 Apr 19. PMID 20403940
- [Background] Guarner F, Bourdet-Sicard R, Brandtzaeg P, Gill HS, McGuirk P, van Eden W, Versalovic J, Weinstock JV, Rook GA. Mechanisms of disease: the hygiene hypothesis revisited. Nat Clin Pract Gastroenterol Hepatol. 2006 May;3(5):275-84. doi: 10.1038/ncpgasthep0471. PMID 16673007
- [Background] Packey CD, Sartor RB. Interplay of commensal and pathogenic bacteria, genetic mutations, and immunoregulatory defects in the pathogenesis of inflammatory bowel diseases. J Intern Med. 2008 Jun;263(6):597-606. doi: 10.1111/j.1365-2796.2008.01962.x. PMID 18479259
- [Background] Macpherson AJ, Harris NL. Interactions between commensal intestinal bacteria and the immune system. Nat Rev Immunol. 2004 Jun;4(6):478-85. doi: 10.1038/nri1373. No abstract available. PMID 15173836
- [Background] Mazmanian SK, Kasper DL. The love-hate relationship between bacterial polysaccharides and the host immune system. Nat Rev Immunol. 2006 Nov;6(11):849-58. doi: 10.1038/nri1956. Epub 2006 Oct 6. PMID 17024229
- [Background] Brooks WA, Santosham M, Naheed A, Goswami D, Wahed MA, Diener-West M, Faruque AS, Black RE. Effect of weekly zinc supplements on incidence of pneumonia and diarrhoea in children younger than 2 years in an urban, low-income population in Bangladesh: randomised controlled trial. Lancet. 2005 Sep 17-23;366(9490):999-1004. doi: 10.1016/S0140-6736(05)67109-7. PMID 16168782
- [Background] Sazawal S, Black RE, Bhan MK, Bhandari N, Sinha A, Jalla S. Zinc supplementation in young children with acute diarrhea in India. N Engl J Med. 1995 Sep 28;333(13):839-44. doi: 10.1056/NEJM199509283331304. PMID 7651474